CLINICAL TRIAL: NCT05917067
Title: Fluorescence Imaging for the Detection and Perfusion of the Parathyroid Glands of Children
Brief Title: Fluorescence Imaging of the Parathyroid Glands of Children
Acronym: FLUOPATCH
Status: Completed | Type: Observational
Sponsor: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Principal Investigator, Daniël van de Berg, MD, MD, Amsterdam UMC, location VUmc
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: 2023.0263
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Childhood Thyroid Gland Carcinoma; Thyroid Diseases
Keywords: Indocyanine Green; ICG-fluorescence angiography; Autofluorescence; Children
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children (<18 years) that will undergo total thyroidectomy for any indication
  Interventions: Diagnostic Test: Fluorescence imaging of the parathyroid glands of children

INTERVENTIONS:
Diagnostic Test: Fluorescence imaging of the parathyroid glands of children — Patients that participate in this study will always receive standard care. For the purpose of this study, the camera settings (i.e. camera distance to the operating field, switching of OR-lights, and angle of the camera on the operating field) and ICG-protocol (i.e. dose, injection speed) will be standardized among the participating centers in order to generate an homogeneous data set for quantification of the fluorescence signal intensity.

SUMMARY:
The aim of this study is to develop a standardized and user-independent imaging workflow model for autofluorescence and quantified fluorescence angiography with Indocyanine Green (ICG) of the parathyroid glands of children. For this purpose, all pediatric patients will undergo thyroid surgery with the use of autofluorescence and quantified ICG-fluorescence.

This study could be the first step in reducing the rate of postoperative hypocalcemia in children, by using fluorescence angiography during pediatric thyroid surgery.

DETAILED DESCRIPTION:
Background:

Children with thyroid cancer have excellent survival rates. However, postoperative hypocalcemia, due to inadvertent excision of the parathyroid glands or damage to their vasculature during thyroid surgery, is a severe complication which occurs in 24% - 67% of the children with thyroid cancer and causes lifelong reduced quality of life and increased morbidity rates. In adults, intraoperative identification of the parathyroid glands with autofluorescence and assessment of their perfusion using quantified ICG-fluorescence angiography has shown to reduce postoperative hypocalcemia. However, in children no studies regarding quantified fluorescence of the parathyroid glands have been conducted. There is a clear need for surgical techniques to identify and preserve the parathyroid glands during thyroid surgery in children.

Therefore, the aim of this study is to develop a standardized imaging workflow model for autofluorescence and quantified ICG-angiography of the parathyroid glands in children. This workflow model can be the first step in reducing the rate of postoperative hypocalcemia in children.

Study design:

This will be a prospective, observational, multicenter, feasibility study. The aim is to generate the patterns of intraoperative autofluorescence and quantified ICG-fluorescence angiography of the parathyroid glands in children, resulting in a user-independent, standardized imaging workflow model for autofluorescence and quantified ICG-angiography of the parathyroid glands of children.

ELIGIBILITY:
Inclusion Criteria:

1. Patients <18 years
2. Patients undergoing total thyroidectomy (for any indication)
3. Patients undergoing lobectomy for the suspicion of a malignancy, with a subsequent completion thyroidectomy
4. Written informed consent (from parents/caregivers, patients or both, see chapter 6.0)

Exclusion Criteria:

1. Patients with preoperative hypo - or hypercalcemia, treated for hypo- or hypercalcemia, (chronic) renal disease, kidney transplantation or any disorder that requires calcium supplementation (other than standard preoperative calcium supplementation for a total thyroidectomy).
2. Patients with known allergy to ICG or iodinated contrast
3. Pregnancy or breastfeeding
4. Patients with severe liver dysfunction
5. Preterm neonates
6. Newborn infants with an indication for exchange transfusion for severe neonatal hyperbilirubinemia

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under 18 years old that will undergo total thyroidectomy for any indication or lobectomy for the suspicion of a malignancy will be checked for the inclusion and excusion criteria. If eligible, patients will be asked for written informed consent.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Number and location of autofluorescent parathyroid glands | During thyroid surgery
  Number and location of autofluorescent parathyroid glands
Quantification of the fluorescent signal of ICG | During thyroid surgery
  Quantification of the fluorescent signal of ICG
Postoperative hypocalcemia | Postoperative day 1-3 and first out-patient clinic visit (between day 1 and day 10 postoperative)
  Postoperative hypocalcemia

OTHER OUTCOMES:
Postoperative calcium supplementation | Postoperative day 1-3 and first out-patient clinic visit (between day 1 and day 10 postoperative)
  Need for (extra) postoperative calcium supplementation
Total duration of the operation | Day of the operation
  Total duration of the operation in minutes
(postoperative) complications, following the Clavien-Dindo classification | During thyroid surgery and day 1-3 till and first out-patient clinic visit (between day 1 and day 10 postoperative)
  Any (postoperative) complications, following the Clavien-Dindo classification
Need for autotransplantation of the parathyroid glands | During thyroid surgery
  Need for autotransplantation of the parathyroid glands by visual assessment (non-fluorescence) of the surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Joep Derikx, MD, PhD, Principal Investigator — Amsterdam UMC - Emma Children's Hospital
Locations (3):
- Netherlands (3):
  - Amsterdam UMC - Emma Children's Hospital, Amsterdam
  - UMC Groningen, Groningen
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Request for data sharing will be considered by the project leaders upon written request. Deidentified participant data will be made available after receipt of a written proposal and a signed data sharing agreement. Furthermore, an amendment will be handed in to the MEC for ethical approval before starting this additional research.
Supporting Information: Study Protocol
Time Frame: The study protocol will be published in a international, peer-reviewed journal with open acces, during the study period.

REFERENCES:
- See also: KiKa funding page for the present study — https://www.kika.nl/onderzoeken-kinderkanker/minder-bijwerkingen-van-operatie-bij-kinderen-met-schildklierkanker